CLINICAL TRIAL: NCT04127266
Title: Expanding Pancreas Donor Pool by Evaluation of Unallocated Organs After Brain Death: The EXPLORE Study
Brief Title: Expanding Pancreas Donor Pool by Evaluation of Unallocated Organs After Brain Death - The EXPLORE Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. A. Mehrabi (Other)
Collaborators: University Hospital Heidelberg (Other); University Hospital Tuebingen (Other); University of Freiburg (Other); Universitätsmedizin Mannheim (Other); German Organ Transplantation Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Dr. A. Mehrabi, Professsor, Head of the Division of Liver Surgery and Visceral Transplantation, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Other Study IDs: S-277/2019
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Unallocated Pancreas Organs
Keywords: Donor pool; Brain death; Unallocated organs; Histopathological quality
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreas graft quality directly affects morbidity and mortality rates after pancreas transplantation (PTx). The criteria for pancreas graft allocation are restricted, which has decreased the number of available organs. Suitable pancreatic allografts are selected based on donor demographics, medical history, and the transplant surgeon's assessment of organ quality during procurement. Quality is assessed based on macroscopic appearance, which is biased by individual experience and personal skills. Therefore, the aim of this study is to assess the histopathological quality of unallocated pancreas organs to determine how many unallocated organs are of suitable quality for PTx, based on histopathologic evaluations. The reasons for allocation rejection will be reported and the correlation between cause of allocation rejection and histopathological quality of the allocated organ will be evaluated.

This is a multicenter cross-sectional explorative study. The demographic data and medical history of donor and cause of rejection of the allocation of graft will be recorded. Organs of included donors will be explanted and macroscopic features such as weight, color, size, and stiffness will be recorded. A tissue sample of the organ will be fixed for further microscopic assessments. Histopathologic assessments will be reported 6 hours (or at time of organ delivery if later than 6 hours), 9 hours, 12 hours, 15 hours, and 18 hours after procurement. 100 pancreases will be evaluated in this study.

DETAILED DESCRIPTION:
With advances in surgery and immunosuppressive therapy, PTx has become an accepted and standardized therapeutic surgery worldwide. Today, PTx is a promising treatment for type 1 diabetes mellitus and for patients undergoing total pancreatectomy because of benign disease. It has been demonstrated that PTx can provide a good glycemic control and insulin independence and improve diabetic lesions including retinopathy, nephropathy, neuropathy, and vasculopathy. Furthermore, thanks to improved immunosuppressive agents, prophylaxis against infections and thrombosis, and modifications in surgical approaches, outcomes after whole organ PTx has consistently improved over the past 20 years. The 1- and 5-year patient survival rates after PTx are approximately 95% and 85%, respectively, and the 1-, and 5-year graft survival rates are 90%, and 70%, respectively.

Morbidity and mortality still occurs after PTx. Morbidity and mortality rates after PTx are mainly related to pancreas graft quality. To decrease these, some restricted criteria for pancreas graft allocation have been defined. However, these allocation criteria have decreased the overall availability of pancreas organs. Consequently, despite an increase in organs from deceased donors, organ utilization (20% of all potential donor pancreases are ultimately used for whole organ transplantation) and also PTx rates (10% overall decline) have decreased. In the US, only 13% of deceased donors provide a pancreas that is utilized for transplantation. Data from Eurotransplant indicate that only 27% of donor pancreases are transplanted, either as whole pancreas grafts or as islet grafts. In addition to the restricted pancreas allocation criteria, some allocated/offered organs are not accepted by transplant surgeons (which is biased by individual experience and personal skills) after an organ quality assessment.

Longer waiting lists, increased waiting times, and donor shortages have increased the need for and number of extended donor criteria organs that are accepted for transplantation. To date, the most important selection criteria to identify suitable pancreatic allografts are donor demographics, donor medical history (age, gender, cause of death, etc.), and the transplant surgeon's own organ quality assessment based on macroscopic appearance. However, it is unclear, whether unallocated organs have a poor histopathologic quality for transplantation. To the best of our knowledge, no systematic histopathologic quality assessment of unallocated pancreas grafts has been performed, so far. In this study, for the first time, the histopathological quality of unallocated pancreas organs from brain-dead donors will be assessed to determine the number of unallocated organs that were potentially suitable for transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible brain-dead organ donors in Baden-Württemberg with consent to donation
* Pancreas reported to Eurotransplant for allocation by the German Organ Transplantation Foundation
* Age ≤ 60 years old
* BMI ≤ 35

Exclusion Criteria:

* Pancreases allocated for transplantation
* Pancreases allocated for islet cell transplantation after being assessed not suitable for solid organ transplantation
* History of pancreas disease
* History of pancreas surgery

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Brain-dead donors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Histopathological quality of pancreas | 18 hours
  Histopathologic features of unallocated organs, including the presence of pancreatitis, fibrosis, edema, hemorragia, steatosis and fat content, dilation of pancreas ducts, and benign/malignant tumors will be reported.

SECONDARY OUTCOMES:
Medical history of donors | One day
Donor Sodium level | One day
  mmol/L
Donor Creatinine level | One day
  mg/dl
Donor Glomerular Filtration rate | One day
Donor Serum Glucose level | One day
  mmol/L
Donor HbA1c rate | One day
Donor Lipase level | One day
  U/l
Donor Amylase level | One day
  U/l
Pre-procurement pancreas allocation suitability score | One day
  Calculated based on age, body mass index, intensive care unit stay, duration of cardiac arrest/asystole, sodium (mmol/L), amylase (U/l), lipase (U/l), inotropic therapy [(nor)adrenaline (γ) or dobuta-/dopamine (γ)].
Macroscopic features of pancreas | One day
  Macroscopic features including stiffness, tissue damage, subscapular hematoma, pancreatic calcification, pancreatic edema, fatty Infiltration, and vascular status.

CONTACTS AND LOCATIONS:
Overall Officials: Arianeb Mehrabi, MD, Principal Investigator — Department of General, Visceral and Transplant Surgery, University Hospital
Locations (1):
- Division of Visceral Transplantation, Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Kulu Y, Khajeh E, Ghamarnejad O, Nikdad M, Sabagh M, Ali-Hasan-Al-Saegh S, Nadalin S, Quante M, Pisarski P, Janigen B, Reissfelder C, Mieth M, Morath C, Goeppert B, Schirmacher P, Strobel O, Hackert T, Zeier M, Springel R, Schleicher C, Buchler MW, Mehrabi A. Expanding pancreas donor pool by evaluation of unallocated organs after brain death: Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Mar;99(10):e19335. doi: 10.1097/MD.0000000000019335. PMID 32150070